CLINICAL TRIAL: NCT02242903
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3079514 in Healthy Subjects
Brief Title: A Study of LY3079514 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 15190; I7B-MC-DPAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3079514 (Experimental): Single dose of LY3079514 administered intravenous (IV) or subcutaneous (SC) during a single occasion
  Interventions: Drug: LY3079514
- Placebo (Placebo Comparator): Single dose of placebo matching LY3079514 administered IV infusion or SC injection during a single occasion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3079514 — Administered SC
  Arms: LY3079514
Drug: LY3079514 — Administered IV
  Arms: LY3079514
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and how well the body will handle a single dose of study drug, LY3079514. This study will last about 12 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants as determined by medical history and physical examination
* To qualify as Japanese for the purpose of this study, the Japanese participant must be first-generation Japanese
* Have a body mass index (BMI) between 18.5 and 32.0 kilograms per square meter (kg/m^2) and have a minimum body weight of 50 kilograms (kg), inclusive at screening
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure that is considered to be clinically significant, as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have known or ongoing psychiatric disorders
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single dose of placebo matching LY3079514 administered intravenous (IV) infusion or subcutaneous (SC) injection during a single occasion.
- LY3079514 Cohort 1: 7 milligrams (mg) single dose of LY3079514 administered by SC injection during a single occasion.
- LY3079514 Cohort 2: 21 mg single dose of LY3079514 administered by SC injection during a single occasion.
- LY3079514 Cohort 3: 70 mg single dose of LY3079514 administered by SC injection during a single occasion.
- LY3079514 Cohort 4: 210 mg single dose of LY3079514 administered by SC injection during a single occasion.
- LY3079514 Cohort 5: 70 mg single dose of LY3079514 administered IV during a single occasion.
- LY3079514 Cohort 6: 210 mg single dose of LY3079514 administered IV during a single occasion.
Period: Overall Study
Arm/Group | Placebo | LY3079514 Cohort 1 | LY3079514 Cohort 2 | LY3079514 Cohort 3 | LY3079514 Cohort 4 | LY3079514 Cohort 5 | LY3079514 Cohort 6
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 11 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LY3079514 (LY) Cohort 1: 7 mg single dose of LY3079514 administered by SC injection during a single occasion
- LY Cohort 2: 21 mg single dose of LY3079514 administered by SC injection during a single occasion
- LY Cohort 3: 70 mg single dose of LY3079514 administered by SC during a single occasion
- LY Cohort 4: 210 mg single dose of LY3079514 administered by SC during a single occasion
- LY Cohort 5: 70 mg single dose of LY3079514 administered IV during a single occasion
- LY Cohort 6: 210 mg single dose of LY3079514 administered IV during a single occasion
- Total: Total of all reporting groups
Arm/Group | Placebo | LY3079514 (LY) Cohort 1 | LY Cohort 2 | LY Cohort 3 | LY Cohort 4 | LY Cohort 5 | LY Cohort 6 | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.96) | 35.5 (10.82) | 34.5 (12.42) | 38.0 (12.82) | 45.3 (12.39) | 39.0 (11.56) | 49.3 (5.61) | 40.5 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 0 | 3 | 0 | 3 | 12
  Male | 8 | 5 | 5 | 6 | 3 | 6 | 3 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 6
  Not Hispanic or Latino | 11 | 6 | 5 | 5 | 5 | 5 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 3 | 0 | 3 | 0 | 3 | 0 | 3 | 12
  Non-Japanese | 9 | 6 | 3 | 6 | 3 | 6 | 3 | 36
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is an adverse event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. A summary of SAEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to Study Completion (Up to 12 Weeks)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | LY3079514 (LY) Cohort 1 | LY Cohort 2 | LY Cohort 3 | LY Cohort 4 | LY Cohort 5 | LY Cohort 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3079514
Time Frame: SC Dosing-Predose,4hr,12hr,24hr,Day(D)3,D5,D8,D11,D15,D22,D29,D43,D57,D85; IV Dosing- D1 and D2 End of Infusion,4hr,12hr,24hr,D3,D8,D15,D22,D29,D36,D43,D57,D85
Population: All randomized participants who received at least 1 dose of study drug and had evaluable Cmax PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- LY Cohort 1: 7 mg single dose of LY3079514 administered by SC injection during a single occasion
- LY Cohort 3: 70 mg single dose of LY3079514 administered by SC injection during a single occasion
- LY Cohort 4: 210 mg single dose of LY3079514 administered by SC injection during a single occasion
Arm/Group | LY Cohort 1 | LY Cohort 2 | LY Cohort 3 | LY Cohort 4 | LY Cohort 5 | LY Cohort 6
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
nanograms/milliliter (ng/mL) | 55.1 (93) | 480 (64) | 3150 (118) | 16900 (45) | 19000 (13) | 41300 (22)

3. Secondary Outcome: PK: Area Under the Concentration Curve Zero to Infinity (AUC 0-∞) of LY3079514
Time Frame: as for outcome 2
Population: All randomized participants who received at least 1 dose of investigational drug and had evaluable AUC PK data. Cohort 1 had zero participants analyzed and was not included in summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram•hour/milliliter (ng•h/mL)
Arm/Group | LY Cohort 1 | LY Cohort 2 | LY Cohort 3 | LY Cohort 4 | LY Cohort 5 | LY Cohort 6
Number analyzed (Participants) | 0 | 4 | 4 | 6 | 6 | 6
nanogram•hour/milliliter (ng•h/mL) |  | 38500 (59) | 402000 (80) | 4850000 (37) | 1240000 (20) | 6470000 (14)

ADVERSE EVENTS:
Arm/Group | Placebo | LY3079514 (LY) Cohort 1 | LY Cohort 2 | LY Cohort 3 | LY Cohort 4 | LY Cohort 5 | LY Cohort 6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/12 | 4/6 | 1/6 | 3/6 | 4/6 | 3/6 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=12) | LY3079514 (LY) Cohort 1 (N=6) | LY Cohort 2 (N=6) | LY Cohort 3 (N=6) | LY Cohort 4 (N=6) | LY Cohort 5 (N=6) | LY Cohort 6 (N=6)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Instillation site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/3 (1) | 0 (0) | 0 (0)
Premenstrual headache (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/3 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days